CLINICAL TRIAL: NCT01497990
Title: Pharmacokinetics of Ertapenem When Used in Empiric Treatment in Burn Patients. Prospective Open Label Study.
Brief Title: Pharmacokinetics Ertapenem Burns
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09/3-W
Record Dates: First submitted 2011-12-15; First posted 2011-12-23 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-11

CONDITIONS: Burn Patients
Keywords: Burns; Ertapenem; Pharmacokinetics
MeSH Terms: conditions — Burns | interventions — Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ertapenem (Experimental): The patient received two injections of ertapenem, at a dose of 1g.j-1 by intravenous injection of 30 minutes, separated by 24 h.
  Interventions: Drug: Ertapenem

INTERVENTIONS:
Drug: Ertapenem — The patient received two injections of ertapenem, at a dose of 1g.j-1 by intravenous injection of 30 minutes, separated by 24 h.

SUMMARY:
This study will examine the pharmacokinetics of ertapenem in ventilated badly (> 30% SCT) burn patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 70 years
* Burned on 30 to 60% of their body surface
* Mechanical ventilation
* Hospitalized in the intensive care unit of Nantes University Hospital for less than 8 days.
* Which the family gave consent
* insured

Exclusion Criteria:

* Patients whose family refused to sign the consent for participation.
* Patients allergic to beta lactam
* Patients with renal failure with creatinine clearance <80 ml.mn-1
* Pregnant women
* Persons protected by the law

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Measurement of serum concentrations of total ertapenem from the second injection in order to calculate Cmax, Vz, ClP , ClR , ClNR , fe, T1/2b et AUC0 - alpha. | Blood samples 5 min after the end of the second injection and 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h after the start of the second injection
  Current study the pharmacokinetics (Cmax, Vz, ClP , ClR , ClNR , fe, T1/2beta, AUC 0 - alpha) in a population of burn patients.

SECONDARY OUTCOMES:
Time between injection and observation of a serum concentration less than the critical concentration below | Blood samples 5 min after the end of the second injection and 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h after the start of the second injection
  Check that the injection of 1 g ertapenem achieves a serum concentration above the critical concentration of bacteria usually isolated in cases of early infection for more than 40% of the time between two injections (t / MIC> 40 %), this ratio being one of the criteria predictive of efficacy of beta-lactam antibiotics.
Time needed between injections in order to obtain a concentration greater than the critical concentration below for the duration of time between two injections | Blood samples 5 min after the end of the second injection and 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h after the start of the second injection
  Study when two injections of ertapenem serum concentrations fall below the critical concentrations of bacteria usually isolated in cases of early infection, if they become.

CONTACTS AND LOCATIONS:
Overall Officials: Ronan LE FLOCH, PH, Study Chair — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France